CLINICAL TRIAL: NCT00917995
Title: STOMAMESH Prospective Randomised Multicenter Trial Concerning the Frequency of Parastomal Hernia With or Without a Mesh
Brief Title: Trial Concerning the Frequency of Parastomal Hernia With or Without a Mesh
Acronym: STOMAMESH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Norrbottens Lans Landsting (Other)
Responsible Party: Principal Investigator, Pia Nasvall, MD, PhD, Norrbottens Lans Landsting
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-081M
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Parastomal Hernia
Keywords: parastomal hernia; prophylactic mesh; colostomy; hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colostomy with a prophylactic mesh (Experimental)
  Interventions: Device: Polypropylene Mesh, density 25-40g/square meter
- Colostomy without a prophylactic mesh (No Intervention)

INTERVENTIONS:
Device: Polypropylene Mesh, density 25-40g/square meter — colostomy with a prophylactic hernia mesh
  Arms: Colostomy with a prophylactic mesh

SUMMARY:
Specific aim:

To compare patients with colostomies with or without mesh at the primary operation. Primary endpoint is the incidence of parastomal hernia requiring surgery.

All patients at participating centers scheduled for permanent colostomy, after signing informed consent and meeting inclusion criteria, will be randomised to formation of a stoma with or without mesh.

If the inclusion criteria is fulfilled and informed consent is signed, the patient is randomised preoperatively.

DETAILED DESCRIPTION:
Parastomal hernia is a relatively common and troublesome complication in patients with a stoma. The exact incidence is not known and depending on definitions and if a bulging is a hernia or not, as well as when after the operation the examination is performed, the incidence varies between 0-48%. A parastomal hernia may give the patient difficulties with appliance and leakage. From an economical point of view a stoma that requires special kinds of appliances is expensive. Theoretically, strengthening of the abdominal wall with a mesh at the the primary operation would reduce the risk for parastomal hernia. Recently presented data suggest that a mesh at the primary operation really does reduce the risk to develop a parastomal hernia. No negative side effects with the use of a mesh have been reported in these studies. All earlier studies have involved relatively small numbers of patients and short times of observation, and therefore under-dimensioned concerning potential negative late side-effects. Complications seen in other studies where mesh has been used in surgery of the bowel include fistulas and infections among others. To understand if mesh at the primary operation, in a safe way, reduces the risk for developing parastomal hernia compared to conventional surgery, is important to perform this new prospective randomised multicenter trial.

Specific aim:

To compare patients with colostomies with or without mesh at the primary operation. Primary endpoint is the incidence of parastomal hernia requiring surgery.

All patients at participating centers scheduled for permanent colostomy, after signing informed consent and meeting inclusion criteria, will be randomised to formation of a stoma with or without mesh.

If the inclusion criteria is fulfilled and informed consent is signed, the patient is randomised preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for permanent colostomy elective or acute operation. The optimal site for stoma is marked preoperatively.
* No previous stoma.
* Over the age of 18.
* Informed consent signed by the patient.

Exclusion Criteria:

* Expected lifetime less then 3 years.
* Fecal peritonitis (perforated bowel with free intestinal content in the peritoneal cavity).
* Previous stoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The number of parastomal hernias in the two groups at 12 and 36 months postoperatively | At 12 and 36 months postoperatively

SECONDARY OUTCOMES:
Quality of life related to health | At 12 and 36 months postoperatively
The health care systems total cost related to the stoma | At 12 and 36 months postoperatively
Rate of infections 30 days postoperatively | At 30 days postoperatively
Late complication related to the mesh leading to surgery | At 12 and 36 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dahlberg, MD PhD, Study Chair — Dept of Surgery Sunderby Hospital, Luela, Sweden
Locations (1):
- Sunderby Hospital, Luleå, Sweden

REFERENCES:
- [Derived] Naverlo S, Gunnarsson U, Strigard K, Nasvall P. Quality of life after end colostomy without mesh and with prophylactic synthetic mesh in sublay position: one-year results of the STOMAMESH trial. Int J Colorectal Dis. 2019 Sep;34(9):1591-1599. doi: 10.1007/s00384-019-03359-2. Epub 2019 Aug 7. PMID 31392405